CLINICAL TRIAL: NCT02745405
Title: Implications of Wearing a Fat Suit for Eating, Physiological Stress, and Psychological Well-Being
Brief Title: Implications of Wearing a Fat Suit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: A. Janet Tomiyama (Other)
Responsible Party: Sponsor-Investigator, A. Janet Tomiyama, Faculty Sponsor, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 13-001873
Record Dates: First submitted 2016-04-11; First posted 2016-04-20 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Feeding Behaviors
Keywords: Weight Stigma; Cortisol Reactivity; Eating Behavior
MeSH Terms: conditions — Feeding Behavior; Weight Prejudice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fat Suit Condition (Experimental): Participants are randomly assigned to wear a fat suit and then walk across campus.
  Interventions: Other: Fat Suit
- Control Condition (Other): Participants are randomly assigned to wear the same clothing that is on the fat suit but in their own size and then walk across campus.
  Interventions: Other: Control Condition

INTERVENTIONS:
Other: Fat Suit — Participants wear a fat suit.
  Arms: Fat Suit Condition
Other: Control Condition — Participants wear same clothing as intervention, but in their own size.
  Arms: Control Condition

SUMMARY:
This study examined how wearing a fat suit might lead individuals to experience the negative effects of weight based stigmatization, including psychological, behavioral, and physiological consequences. It also aimed to test using the fat suit as a possible intervention tactic to reduce weight stigma.

DETAILED DESCRIPTION:
The goal of this study was to understand how embodying a stigmatized domain might elicit the same consequences investigators see in victims of weight stigma. Participants were randomly assigned to either manipulate their weight through wearing a fat suit prosthesis or to a control condition where they wore the same clothing that was on the fat suit but in their own size. Outcome variables were cortisol reactivity, psychological well-being, and food and drink consumption. Additionally, this study tested whether wearing the fat suit might serve as an effective weight stigma reduction effort.

ELIGIBILITY:
Inclusion Criteria:

* Participants had to be registered in the UCLA Department of Psychology Subject Pool.

Exclusion Criteria:

* No specific exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2014-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Eating behavior measured via grams of food consumed | ~10-minutes post-manipulation
  M&Ms, potato chips, and full-sugar soda consumption

SECONDARY OUTCOMES:
Cortisol reactivity | ~20 minutes post-manipulation
Antifat Attitudes measured via electronic questionnaire | ~30 minutes after post-manipulation
Psychological Well-Being measured via electronic questionnaires | ~15 minutes post-manipulation

CONTACTS AND LOCATIONS:
Overall Officials: A. Janet Tomiyama, Ph.D, Principal Investigator — University of California, Los Angeles

IPD SHARING:
Plan to Share IPD: Undecided
Interested individuals should contact the PI, who will consult with the UCLA IRB regarding the request.

REFERENCES:
- [Background] Crandall CS. Prejudice against fat people: ideology and self-interest. J Pers Soc Psychol. 1994 May;66(5):882-94. doi: 10.1037//0022-3514.66.5.882. PMID 8014833
- [Background] Baker F, Denniston M, Zabora J, Polland A, Dudley WN. A POMS short form for cancer patients: psychometric and structural evaluation. Psychooncology. 2002 Jul-Aug;11(4):273-81. doi: 10.1002/pon.564. PMID 12203741
- [Background] Zadro L, Williams KD, Richardson R. How low can you go? Ostracism by a computer is sufficient to lower self-reported levels of belonging, control, self-esteem, and meaningful existence. Journal of Experimental Social Psychology, 40(4): 560-567, 2004.
- [Derived] Incollingo Rodriguez AC, Heldreth CM, Tomiyama AJ. Putting on weight stigma: A randomized study of the effects of wearing a fat suit on eating, well-being, and cortisol. Obesity (Silver Spring). 2016 Sep;24(9):1892-8. doi: 10.1002/oby.21575. Epub 2016 Jul 28. PMID 27465666